CLINICAL TRIAL: NCT01677273
Title: The Effect of Hydrolyzed Casein on Energy Expenditure and Subjective Appetite
Acronym: HerKulES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Arla Foods (Industry); The Danish Dairy Research Foundation, Denmark (Other); FrieslandCampina (Industry)
Responsible Party: Principal Investigator, AAstrup, Prof., MD, Head of Department, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: B299
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Increased Energy Expenditure; Increased Satiety
Keywords: Respiratory chambers; Energy expenditure; Appetite; Dairy proteins; Diet induced thermogenesis; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydrolyzed casein (Active Comparator): Hydrolyzed casein
  Interventions: Dietary Supplement: Hydrolyzed casein
- Intact casein (Active Comparator): Intact casein
  Interventions: Dietary Supplement: Intact casein
- Intact whey protein (Active Comparator): Intact whey protein
  Interventions: Dietary Supplement: Intact whey protein

INTERVENTIONS:
Dietary Supplement: Hydrolyzed casein — 30 g protein/supplement, 4 supplements/visit
  Other Names: Hyvital casein CMA 500, Friesland Campina
  Arms: Hydrolyzed casein
Dietary Supplement: Intact casein — 30 g protein/supplement, 4 supplements/visit
  Other Names: Miprodan 30, Arla Foods
  Arms: Intact casein
Dietary Supplement: Intact whey protein — 30 g protein/supplement, 4 supplements/visit
  Other Names: Lacprodan SP-9225 Instant, Arla Foods
  Arms: Intact whey protein

SUMMARY:
The primary aim is to examine and compare the effects of hydrolyzed casein (HC), intact casein (IC) and intact whey protein (IWP) on diet-induced thermogenesis (DIT). Furthermore, to study the effects on appetite regulation assessed by subjective appetite sensations, ad libitum energy intake and appetite regulating hormones.

Whey and casein differ in absorption and digestion rate, with whey being a fast protein and casein being a slow protein. When casein undergoes hydrolysis the absorption and digestion rates approaches the rates of whey. In the present study the importance of absorption rate and amino acid composition, in regards to energy expenditure and appetite regulation, will be examined. HC and IC have identical amino acid composition, but differ in absorption rate, whereas HC and IWP have similar absorption rates, but differ in amino acid composition. We hypothesize that consumption of HC will increase DIT and fat oxidation to a greater extend that IC. Moreover, that HC and IWP will increase satiety shortly after protein consumption, whereas IC will be more satiating after several hours.

The study is a controlled, randomized, 3-arm crossover study. It consists of three visits in a respiratory chamber separated by at least two weeks. 26 healthy, overweight and obese (BMI 27-35 kg/m2) young men will be enrolled and randomized to the order of the three protein supplements (HC, IC or IWP). At each visit protein supplements (containing either HC, IC or IWP) will be served as breakfast, lunch and dinner. Respiratory measures will be obtained over 24 hours and appetite will be assessed by visual analogue scales and appetite regulating hormones. Furthermore, ad libitum energy intake will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men and woman
* Overweight and obese (BMI 27-35 kg/m2)
* 18-40 years
* Women must have a regular menstrual cycle

Exclusion Criteria:

* Allergic to dairy products or other food components
* Vegetarians
* Weight change >3kg within 2 months prior to start of the study
* Use of alcohol >14 drinks/wk
* Drug abuse
* Smoking
* Physically active >10 hrs/wk
* Use of over-the-counter or prescription medication that influences body weight, appetite or metabolism
* Diabetes Mellitus
* Dyslipidemia
* Diseases, which influence metabolism
* Donation of blood 3 months prior to start of the study
* Subjects with a hemoglobin value < 8 mol/L (measured at screening)
* Subjects with a blood glucose level > 6.1 mmol/l (110 mg/dl) (measured at screening)
* Subjects who are unable to give an informed consent.
* Pregnant and lactating women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Diet-induced thermogenesis | 24 hours

SECONDARY OUTCOMES:
Appetite assessed by visual analogue scales | 24 hours
Appetite assessed by ad libitum energy intake | 1 single meal
Appetite regulating hormones in plasma | 4 hours
Components of respiratory measures (basal metabolic rate, sleeping metabolic rate and substrate oxidations) | 24 hours
Differences in insulin, glucose and atrial natriuretic peptide | 4 hours
Ad libitum energy intake assessed by 24 hour dietary records | 24 hours
NMR-spectroscopy based metabonomics profiling of urin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof., MD, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen
Locations (1):
- Department of Human Nutrion, Frederiksberg, Denmark